CLINICAL TRIAL: NCT02137369
Title: Testing an Imaging Biomarker for Treatment Stratification in Major Depression
Brief Title: The ISLAND Study: InSuLa Assessed Needs for Depression
Acronym: ISLAND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Boadie W. Dunlop, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00073702; R01MH073719 (NIH); 00073702 (Other: Emory)
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Depression
Keywords: MDD; Major Depressive Disorder; Treatment; Antidepressants; Lexapro; Talk therapy
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Escitalopram; Sertraline; Antidepressive Agents; Cognitive Behavioral Therapy; Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SSRI (Active Comparator): Escitalopram, pill form, 20mg-40mg, daily, for 12 weeks or Sertraline, pill form, 50 - 150 mg, daily for 12 weeks
  Interventions: Drug: Selective serotonin re-uptake inhibitor; Other: Combination treatment (SSRI + CBT)
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy (CBT) CBT will include 16 1-hour sessions provided over 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Other: Combination treatment (SSRI + CBT)

INTERVENTIONS:
Drug: Selective serotonin re-uptake inhibitor — Escitalopram, 20mg-40mg daily or Sertraline 50-150 mg daily for 12 weeks
  Other Names: Escitalopram or Sertraline; SSRI; Antidepressant medication; Depression treatment
  Arms: SSRI
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy, standardized, 16 sessions over 12 weeks.
  Other Names: CBT; Depression Treatment; Talk therapy
  Arms: Cognitive Behavioral Therapy
Other: Combination treatment (SSRI + CBT) — study participants who do not remit in the first 12 weeks will be offered combination treatment of both treatments for 12 more weeks.
  Other Names: Crossover treatment; escitalopram; depression treatment; antidepressant; talk therapy; depression trial

SUMMARY:
While there are many effective options for treating a major depressive episode, there are no clinical markers that predict the likelihood of remission with an initial trial of either an antidepressant medication or psychotherapy. The goal of this study is to test how brain function changes in depress patients treated with cognitive behavioral therapy (CBT) compared to patients treated with a selective serotonin reuptake inhibitor (SSRI, either escitalopram or sertraline), which are FDA approved antidepressants. The study aims to determine if bran scan findings might help physicians to select the most effective antidepressant treatment for an individual patient.

Up to 100 male and female outpatients who are between 21-55 years old will be enrolled. Participation in the study will last from 14-26 weeks.

Subjects will be randomized to receive either escitalopram (s-CIT) or CBT for 12 weeks. Resting-state positron emission tomography (PET) and BOLD functional magnetic resonance imaging (fMRI) scans will be done before the treatment begins, and again at the end of treatment (week 12). Non-responders to s-cIT or CBT will be crossed over to receive an additional 12 weeks of treatment with the alternative intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 18-60 years.
2. Primary psychiatric diagnosis of Major Depressive Disorder, without psychotic features, confirmed via SCID-IV structured diagnostic interview.
3. Screening Hamilton Depression Rating Scale (HAMD) ≥ 18; and Baseline HAMD ≥ 15.
4. If the patient is a woman of child-bearing potential, she must agree to use an acceptable form of birth control for duration of study participation.
5. Able to understand and provide informed consent for participation.

Exclusion Criteria:

1. Lifetime history of Bipolar Disorder, Dementia, Autism Spectrum Disorder, Schizophrenia, or any other Psychotic Disorder.
2. Psychotic symptoms occurring at any time during the current major depressive episode.
3. Current (past 12 months) diagnosis of Panic disorder, Obsessive Compulsive Disorder, Posttraumatic Stress Disorder, Anorexia Nervosa, or Bulimia Nervosa.
4. Alcohol or Drug Dependence within 12 months or Abuse within 3 months (excluding nicotine and caffeine) of baseline visit, as assessed by history and urine drug screen.
5. Clinical evidence of a severe Personality Disorder, as assessed by the study psychiatrist, which would impede participation or completion of the trial.
6. Known neurological disorders or documented serious head injury.
7. Serious and unstable medical illnesses including cardiovascular disease and cancer.
8. Active medical conditions with known mood changes (endocrine, autoimmune disorders).
9. Current diabetes mellitus.
10. For women, pregnancy, lactation, or unwillingness to comply with birth control requirements.
11. Use of any of the following treatments or any other alternative therapy within 2 weeks of the pre-treatment PET scan that may have beneficial effects on mood, including St John's Wort, S-adenosyl methionine (SAMe), n-3 fatty acids, or light therapy.
12. Use of antidepressant medication within 1 month of the pre-treatment PET scan (within 5 weeks for fluoxetine and protryptyline).
13. Failure to achieve a much improved status (i.e. equivalent to >50% symptom reduction) with 1) any lifetime treatment course of CBT (defined as a minimum of 4 sessions of a specified manual-driven therapy by a CBT-trained therapist) or 2) both escitalopram and sertraline (defined as a minimum of 6 weeks of at the minimum effective dose).
14. Clinically significant active suicidal ideation or self-injurious behavior necessitating immediate treatment, as determined by the investigator.
15. Received electroconvulsive therapy in the past 6 months or during the current depressive episode.
16. Currently responding to medication treatment, without clinical reasons to change.
17. Current treatment with weekly individual or group psychotherapy of any type targeted at depressive symptoms.
18. QTc >500 milliseconds on EKG at screening.
19. Contraindications for MRI, including, but not limited to pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, intra-uterine devices for birth control.
20. Use of concomitant medications with the exception of:

    * Maintenance or prophylactic therapy for stable medical conditions.
    * Hypnotic medication prescribed or approved by the study physician, (up to a three doses per week) for insomnia, as long if not the night before a PET/MRI or clinic ratings visit. Antipsychotic medications, whether prescribed for sleep or other indications, are prohibited.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2014-09; Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boadie W Dunlop, MD/MS, Principal Investigator — Emory University
Locations (1):
- 12 Executive Park Drive, 3rd floor, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Kelley ME, Choi KS, Rajendra JK, Craighead WE, Rakofsky JJ, Dunlop BW, Mayberg HS. Establishing Evidence for Clinical Utility of a Neuroimaging Biomarker in Major Depressive Disorder: Prospective Testing and Implementation Challenges. Biol Psychiatry. 2021 Aug 15;90(4):236-242. doi: 10.1016/j.biopsych.2021.02.966. Epub 2021 Feb 26. PMID 33896622
- See also: Study information — http://www.emoryclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 77 were consented, 60 started treatments
Groups:
- SSRI: Escitalopram, pill form, 20mg-40mg, daily, for 12 weeks OR Sertraline, pill form, 50-150 mg, daily for 12 weeks.
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy (CBT)
  Cognitive Behavioral Therapy: Cognitive Behavioral Therapy, standardized, 16 1-hour sessions over 12 weeks.
Period: Overall Study
Arm/Group | SSRI | Cognitive Behavioral Therapy
Started | 49 | 11
Completed | 41 | 9
Not Completed | 8 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Moved away | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- SSRI: Escitalopram, pill form, 20mg-40mg, daily, for 12 weeks OR Sertraline, pill form, 50-150 mg, daily, for 12 weeks
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy (CBT) CBT will include 16 1-hour standardized sessions provided over 12 weeks.
- Total: Total of all reporting groups
Arm/Group | SSRI | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 49 | 11 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 11 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 8 | 43
  Male | 14 | 3 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 28 | 6 | 34
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 49 | 11 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Remission From Major Depressive Episode Events
Description: Remission from major depressive episode as assessed by 17-item Hamilton Depression Rating Scale.
Time Frame: 12 weeks
Measure: Number; unit: number of events
Groups:
- SSRI: Escitalopram, pill form, 20mg-40mg, daily, for 12 weeks, OR
  Sertraline, [pill form, 50-150 mg, daily for 12 weeks
Arm/Group | SSRI | Cognitive Behavioral Therapy
Number analyzed (Participants) | 49 | 11
number of events | 15 | 4

2. Secondary Outcome: Number of Response to Treatment Events
Description: Response Defined as 50% Change in Hamilton Depression Rating Scale-17 Score at 12 Weeks
Time Frame: 12 weeks
Measure: Number; unit: number of events
Groups:
- SSRI: Escitalopram, pill form, 20mg-40mg, daily, for 12 weeks, OR Sertraline, pill form, 50-150 mg, daily, for 12 weeks
Arm/Group | SSRI | Cognitive Behavioral Therapy
Number analyzed (Participants) | 49 | 11
number of events | 21 | 5

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | SSRI | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/11
Other Adverse Events (participants affected / at risk) | 44/49 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSRI (N=49) | Cognitive Behavioral Therapy (N=11)
Hospitalization for suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSRI (N=49) | Cognitive Behavioral Therapy (N=11)
Headache (General disorders) | 19 (21) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (13) | 0 (0)
Insomnia (Nervous system disorders) | 9 (10) | 0 (0)
Diarea (Gastrointestinal disorders) | 8 (9) | 0 (0)
Anxiety (Psychiatric disorders) | 9 (9) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1)
Sedation (Surgical and medical procedures) | 8 (8) | 1 (1)
Reduced Concentration (General disorders) | 7 (7) | 0 (0)
Fatigue (General disorders) | 7 (7) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 0 (0)
Libido reduced (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Restlessness (Nervous system disorders) | 4 (4) | 0 (0)
Paresthesia (Nervous system disorders) | 4 (4) | 0 (0)
Sweating (General disorders) | 4 (4) | 0 (0)
Yawning (General disorders) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Abnormal Dreams (Nervous system disorders) | 3 (3) | 0 (0)
Reduced Appetite (General disorders) | 3 (3) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Blurred vision (Eye disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 0 (0)
Abdominal pain (General disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dry mouth (General disorders) | 2 (2) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cognitive slowing (Psychiatric disorders) | 1 (1) | 0 (0)
Increased Appetite (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Myoclonic jerks (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional blunting (Psychiatric disorders) | 1 (1) | 0 (0)
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Orgasm abnormal (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0)
Weight gain (General disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Mouth Sores (Infections and infestations) | 1 (1) | 0 (0)
Bacterial vaginosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Difficulty swallowing (General disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Worsening depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal calculus (Renal and urinary disorders) | 1 (1) | 0 (0)
Jaw tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased Urination (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT02137369/Prot_SAP_000.pdf